CLINICAL TRIAL: NCT06342973
Title: Horizontal Ridge Augmentation With Demineralized Bone Allograft Layered With Xenograft - a Prospective Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Geistlich Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5591
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-06

CONDITIONS: Alveolar Ridge Deficiency
Keywords: Horizontal ridge augmentation; Bone atrophy; Bone graft; Dental implant
MeSH Terms: interventions — Transplantation, Heterologous; Transplantation, Homologous

STUDY DESIGN:
Intervention Model Description: Single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Xenograft and allograft (Experimental): The group will consist of patients receiving horizontal ridge augmentation using a combination of Demineralized Freeze Dried Bone Allograft (DFDBA) layered with xenograft particulate bone using a resorbable collagen membrane. The DFDBA will be used internally in contact with the native bone and xenograft will be layered buccal to it.
  Interventions: Device: Xenograft and allograft

INTERVENTIONS:
Device: Xenograft and allograft — For the guided bone augmentation procedure, a crestal incision with one or two vertical incision will be made and a full thickness mucoperiosteal flap will be elevated. Decortication will be performed and the patient will receive grafting with DFDBA with a buccal overlay of xenograft. A bi-layered native collagen membrane will be used and fixed with tacks or sutures. Periosteal incisions will be made to get tension free primary closure. The flap will be closed with sutures. Patients will be prescribed antibiotics, analgesics and mouth rinses as appropriate.

SUMMARY:
The aim of this case series is to evaluate the outcomes of horizontal ridge augmentation performed using a combination of demineralized freeze-dried bone allograft layered with xenograft bone with a resorbable native collagen membrane.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the outcomes of horizontal gone gain when demineralized freeze dried bone allograft (DFDBA) and xenograft are used in a layering technique.

Primary objectives are to compare the bone gain after the bone augmentation procedure. Secondary outcomes are to study the vital bone percentage formation after the bone augmentation procedure and to study the amount of shrinkage of the graft material observed after the procedure.

Test group will consist of patients receiving horizontal ridge augmentation using a combination of DFDBA layered with xenograft particulate bone using a resorbable collagen membrane. Surgical procedure is describe under assigned interventions.

Follow up and implant placement:

The patients will be followed up at 1-2, 3-5 and 6-8 weeks to assess the surgical site for healing. Following this, the patient will be allowed to heal for a period of 6-9 months at which point a cone beam computed tomography (CBCT) will be taken to evaluate the bone gain after horizontal ridge augmentation.

CBCT Measurements:

The images obtained from the CBCT scan will be transferred to a digital CBCT viewing software in which measurements will be carried out. The anatomical landmarks and adjacent teeth will be identified and used to orient the scan to get an image representing the buccal-palatal plane of the area of interest. The horizontal bone gain will be measured at 3,5,7 mm from the crest. Additionally, the amount of graft shrinkage will be measured between immediate post-operative CBCT and follow up CBCT.

Bone core biopsies:

Following at least 6 months of healing and follow up, patients will be appointed for implant placement. At this visit a full thickness flap will be raised. If anatomical considerations and space permits, a bone core biopsy will be obtained using a trephine and stored in formalin for histologic and histo-morphometric analysis. The harvesting of a bone core is considered additional for the study. It will only be performed if it is safe to do so and the harvesting of the core will not jeopardize the long-term longevity of the implant placement (not all patients that are part of the study will undergo the harvesting of a bone core). This bone core will be saved for histologic analysis.

Histologic preparation and evaluation:

Following the bone core removal, the biopsied specimens will be stored until further evaluation. The bone core biopsies will be prepared and evaluated at a lab. De-identified samples will be shipped to the lab for further analysis. Briefly, the biopsy will be dehydrated in a series of ethanol baths. Following this, it will be infiltrated in xylene and methyl metha-acrylate. Following embedding, the bone samples will be sectioned using a hard tissue microtome and stained with hematoxylin-eosin. The quantitative assessment of percentage vital bone, graft particles and connective tissue will be measured using a grid under magnification.

ELIGIBILITY:
Inclusion Criteria:

Patients at least 18 years of age Patients requiring horizontal bone augmentation prior to implant placement ASA I or ASA II patients Non-smoker Patients willing to be followed up for a period of 6-9 months Patients must be physically able to tolerate conventional surgical procedure or procedures under IV moderate sedation.

Exclusion Criteria:

Patients with uncontrolled diabetes Patients with history of radiation to the jaw Patient with immune compromise due to disease or medication Patients requiring primarily vertical bone augmentation prior to implant placement Patients taking bisphosphonates Patients with HIV or hepatitis infection Patients who are known to be pregnant or planning to within 6 months of study enrollment Patients with a history of a failed implant in the site. Patients with an active infection or pathology in the site of treatment that need to be treated prior to bone augmentation Patients with a history of untreated generalized chronic periodontitis Patients who are unable to provide consent and require a legally authorized representative to sign on their behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Amount of horizontal bone gain | 6-9 months
  Horizontal bone gain will be measured from post operative CBCT scans taken 6-9 months following the procedure
Percentage of Vital bone | 6-9 months
  Vital bone percentage will be measured from the bone core trephines taken 6-9 months after the procedure during implant placement
Amount of graft shrinkage | 6-9 months
  Graft shrinkage will be measured as the change in horizontal bone width between immediate post operative CBCT scans and scans taken at 6-9 months

SECONDARY OUTCOMES:
Incidence of surgical complications | 1-2 weeks, 3-5 weeks, 6-8 weeks
  Surgical complications will be noted during the healing period

CONTACTS AND LOCATIONS:
Overall Officials: Eswar Kandaswamy, MS, Principal Investigator — LSUHSC School of Dentistry
Locations (1):
- LSUHSC School of Dentistry, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No